CLINICAL TRIAL: NCT00701038
Title: The Role of Diagnosis and Treatment of Sleep Apnea in the Acute Exacerbation of Heart Failure
Brief Title: Diagnosis and Treatment of Sleep Apnea in the Acute Exacerbation of Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rami Khayat (Other)
Responsible Party: Sponsor-Investigator, Rami Khayat, Associate Professor-Clinical, Ohio State University
Organization: Ohio State University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2005H0186
Record Dates: First submitted 2008-06-17; First posted 2008-06-19 (Estimated); Results first posted 2011-12-14 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2013-01

CONDITIONS: Sleep Apnea; Heart Failure
Keywords: Sleep apnea,; obstructive sleep apnea,; heart failure,; CHF
MeSH Terms: conditions — Sleep Apnea Syndromes; Heart Failure; Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Device (Experimental): Provided with an auto adjusting bi-level positive airway pressure device
  Interventions: Device: auto adjusting bi-level positive airway pressure device
- Control (No Intervention): No device

INTERVENTIONS:
Device: auto adjusting bi-level positive airway pressure device — auto adjusting bi-level positive airway pressure device is provided for treatment of obstructive sleep apnea.
  Other Names: APAP; CPAP
  Arms: Device

SUMMARY:
Congestive heart failure affects 2.3 percent of the population (approximately 4,900,000) with an incidence of 10 per 1,000 of the population after the age of 65 (1). The admission rate for patients with heart failure is on the rise, so is the mortality associated with it and its national annual bill, now exceeding $21 billion (1). Obstructive Sleep Apnea (OSA) is present in 11-37 percent of patients with heart failure (2,3), and tends to increase in severity when the heart failure is less controlled (4, 5). Therefore, the actual prevalence of OSA in patients hospitalized with acute heart failure is likely higher. There is now evidence that treatment of OSA with nasal Continuous Positive Pressure (nCPAP) in outpatients with stable heart failure improves left ventricular ejection fraction, and quality of life (6), and confers a reduction in fatal and non-fatal cardiovascular events (7). However, there has not been any evaluation of the role of diagnosis and treatment of OSA in patients hospitalized with acute heart failure. This uncertainty about the true prevalence and role of OSA in exacerbations of heart failure, and the role of its treatment in the acute setting may explain why aggressive diagnostic and therapeutic strategy for OSA in patients admitted to the hospital with acute heart failure is not part of the standard clinical practice in acute care centers. Given the rising admission rate, and mortality associated with heart failure, an evaluation of the role of OSA and its treatment in this patient population is highly significant.

DETAILED DESCRIPTION:
OSA is associated with large negative swings in the intrathoracic pressure, significant increase in the sympathetic nerve activity and repetitive surges in blood pressure, along with episodic hypoxia and hypercapnea (8, 9). These autonomic and respiratory changes may increase the cardiac muscle workload, cardiac dysrrhythmia, and exacerbate ischemia (10,11,12). Treatment with continuous positive airway pressure (CPAP) is the most successful therapeutic modality available for obstructive sleep apnea. It is still not clear whether establishing the diagnosis of OSA and initiating treatment with CPAP while still in the hospital carries any benefit in the management of patients with acute heart failure. This study will evaluate the effect of work up and treatment of OSA on the outcome of patients hospitalized with acute congestive heart failure (CHF).

ELIGIBILITY:
.Inclusion Criteria:

* Able to provide an informed consent
* Speaks English
* Older than 21
* Heart Failure
* Positive for OSA

Exclusion Criteria:

* CSA
* Already on CPAP
* Hemodynamic instability
* Acute respiratory failure
* Neurological defect
* Dialysis

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2006-08; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rami N Khayat, MD, Principal Investigator — Ohio State University

REFERENCES:
- [Background] Heart Disease and Stroke-Statistics, American Heart Association, 2005 update
- [Background] Javaheri S, Parker TJ, Liming JD, Corbett WS, Nishiyama H, Wexler L, Roselle GA. Sleep apnea in 81 ambulatory male patients with stable heart failure. Types and their prevalences, consequences, and presentations. Circulation. 1998 Jun 2;97(21):2154-9. doi: 10.1161/01.cir.97.21.2154. PMID 9626176
- [Background] Sin DD, Fitzgerald F, Parker JD, Newton G, Floras JS, Bradley TD. Risk factors for central and obstructive sleep apnea in 450 men and women with congestive heart failure. Am J Respir Crit Care Med. 1999 Oct;160(4):1101-6. doi: 10.1164/ajrccm.160.4.9903020. PMID 10508793
- [Background] Skinner MA, Choudhury MS, Homan SD, Cowan JO, Wilkins GT, Taylor DR. Accuracy of monitoring for sleep-related breathing disorders in the coronary care unit. Chest. 2005 Jan;127(1):66-71. doi: 10.1378/chest.127.1.66. PMID 15653964
- [Background] Solin P, Bergin P, Richardson M, Kaye DM, Walters EH, Naughton MT. Influence of pulmonary capillary wedge pressure on central apnea in heart failure. Circulation. 1999 Mar 30;99(12):1574-9. doi: 10.1161/01.cir.99.12.1574. PMID 10096933
- [Background] Mansfield DR, Gollogly NC, Kaye DM, Richardson M, Bergin P, Naughton MT. Controlled trial of continuous positive airway pressure in obstructive sleep apnea and heart failure. Am J Respir Crit Care Med. 2004 Feb 1;169(3):361-6. doi: 10.1164/rccm.200306-752OC. Epub 2003 Nov 3. PMID 14597482
- [Background] Marin JM, Carrizo SJ, Vicente E, Agusti AG. Long-term cardiovascular outcomes in men with obstructive sleep apnoea-hypopnoea with or without treatment with continuous positive airway pressure: an observational study. Lancet. 2005 Mar 19-25;365(9464):1046-53. doi: 10.1016/S0140-6736(05)71141-7. PMID 15781100
- [Background] Katragadda S, Xie A, Puleo D, Skatrud JB, Morgan BJ. Neural mechanism of the pressor response to obstructive and nonobstructive apnea. J Appl Physiol (1985). 1997 Dec;83(6):2048-54. doi: 10.1152/jappl.1997.83.6.2048. PMID 9390980
- [Background] Morgan BJ, Denahan T, Ebert TJ. Neurocirculatory consequences of negative intrathoracic pressure vs. asphyxia during voluntary apnea. J Appl Physiol (1985). 1993 Jun;74(6):2969-75. doi: 10.1152/jappl.1993.74.6.2969. PMID 8365996
- [Background] Magder SA, Lichtenstein S, Adelman AG. Effect of negative pleural pressure on left ventricular hemodynamics. Am J Cardiol. 1983 Sep 1;52(5):588-93. doi: 10.1016/0002-9149(83)90032-2. PMID 6613883
- [Background] Stoohs R, Guilleminault C. Cardiovascular changes associated with obstructive sleep apnea syndrome. J Appl Physiol (1985). 1992 Feb;72(2):583-9. doi: 10.1152/jappl.1992.72.2.583. PMID 1559936
- [Background] Hanly P, Sasson Z, Zuberi N, Lunn K. ST-segment depression during sleep in obstructive sleep apnea. Am J Cardiol. 1993 Jun 1;71(15):1341-5. doi: 10.1016/0002-9149(93)90552-n. PMID 8498378
- [Background] Roebuck T, Solin P, Kaye DM, Bergin P, Bailey M, Naughton MT. Increased long-term mortality in heart failure due to sleep apnoea is not yet proven. Eur Respir J. 2004 May;23(5):735-40. doi: 10.1183/09031936.04.00060404. PMID 15176689
- [Derived] Khayat RN, Abraham WT, Patt B, Pu M, Jarjoura D. In-hospital treatment of obstructive sleep apnea during decompensation of heart failure. Chest. 2009 Oct;136(4):991-997. doi: 10.1378/chest.09-0597. Epub 2009 Jun 30. PMID 19567491

RESULTS

PARTICIPANT FLOW:
Groups:
- Device: Provided with an auto adjusting bi-level positive airway pressure device for 3 days in hospital
- Control: No auto adjusting bi-level positive airway pressure device given during hospital stay
Period: Overall Study
Arm/Group | Device | Control
Started | 27 | 27
Completed | 23 | 23
Not Completed | 4 | 4
Not completed — study amended pilot group of patients | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Device | Control | Total
Number analyzed (Participants) | 27 | 27 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 14 | 37
  >=65 years | 4 | 13 | 17
Age Continuous [Mean (Standard Deviation); unit: years] | 62 (14) | 51 (12) | 56 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 20 | 19 | 39
Region of Enrollment [Number; unit: participants]
  United States | 27 | 27 | 54

OUTCOME MEASURES:

1. Primary Outcome: Left Ventricular Ejection Fraction Improvement
Description: Left ventricular function was assessed using doppler ultrasound. Positive increase in left ventricular function from baseline to 3 nights post treatment indicates potential beneficial impact of treatment on heart function.
Time Frame: baseline and again after three nights in hospital
Population: ITT
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Device | Control
Number analyzed (Participants) | 23 | 23
percent change | 4.5 (1.7) | -.3 (1.5)

ADVERSE EVENTS:
Arm/Group | Device | Control
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 0/27 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No